CLINICAL TRIAL: NCT05088681
Title: Synergic Control of Posture in Peripheral Neuropathies' Patients
Acronym: NEUPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: NEUPER
Record Dates: First submitted 2021-09-11; First posted 2021-10-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Neuropathies
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripheral neuropathies patients: Peripheral neuropathies patients will be assessed at baseline, after a 20 session 2-3/w program of physical therapy and at a follow up of 3 months with:
  * Total Neuropathy Score-clinical version (TNSc©)
  * Nerve conduction studies
  * Short Form Health Survey 36 (SF-36)
  * Functional Independence Measure (FIM)
  * postural evaluation recording during three different postural tasks (quiet standing, voluntary sway and shoulder flexion):centre of pressure (COP) displacement of force platform; surface muscle activation using electromyography (EMG) of 13 muscle on the right side of the body (tibialis anterior, soleus,gastrocnemius lateralis-medialis, biceps femoris, semitendinosus, rectus femoris, vastus lateralis and medialis, tensor fasciae latae, lumbar and thoracic erector spinae and rectus abdominis)
  * Six Minute Walking Test (6MWT), Mini Balance Evaluation System Test (MiniBESTest) and Timed Up and Go test (TUG).
  Interventions: Other: Rehabilitation program
- Healthy age-matched subjects: Healthy age-matched subjects will receive a postural evaluation recording during three different postural tasks (quiet standing, voluntary sway and shoulder flexion):
  * centre of pressure (COP) displacement of force platform;
  * surface muscle activation using electromyography (EMG) of 13 muscle on the right side of the body (tibialis anterior, soleus,gastrocnemius lateralis-medialis, biceps femoris, semitendinosus, rectus femoris, vastus lateralis and medialis, tensor fasciae latae, lumbar and thoracic erector spinae and rectus abdominis).

INTERVENTIONS:
Other: Rehabilitation program — The exercise intervention will consist of an individualized prescription of resistance training, balance training and cardiovascular exercises delivered for 20 session, one-hour, two/three times per week.
  Groups: Peripheral neuropathies patients

SUMMARY:
This is a multicenter observational study aimed to characterize multi-muscle synergy organization in relation to postural stability in individuals with Peripheral Neuropathies (PN) compared to healthy age-matched subjects and to assess the effectiveness of a rehabilitation program driven by multi-muscle synergy organization.

DETAILED DESCRIPTION:
This is a multicenter observational study of peripheral neuropathies patients aiming at characterizing multi-muscle synergy and at assessing the effectiveness of a rehabilitation program driven by multi-muscle synergy organization.

The study can be divided in two phases:

Phase 1 will included peripheral neuropathies patients and healthy age-matched subjects.

Peripheral neuropathies patients will be assessed with:

* Neurological assessment formalized via Total Neuropathy Score-clinical version (TNSc©)
* Nerve conduction studies
* Impact of PN on patients' quality of life using Short Form Health Survey 36 (SF-36)
* Functional status using Functional Independence Measure (FIM)

Peripheral neuropathies patients and healthy age-matched subjects will receive a postural evaluation recording during three different postural tasks (quiet standing, voluntary sway and shoulder flexion):

* centre of pressure (COP) displacement of force platform;
* surface muscle activation using electromyography (EMG) of 13 muscle on the right side of the body (tibialis anterior, soleus,gastrocnemius lateralis-medialis, biceps femoris, semitendinosus, rectus femoris, vastus lateralis and medialis, tensor fasciae latae, lumbar and thoracic erector spinae and rectus abdominis).

Phase 2 will included only peripheral neuropathies patients. Participants will be assessed at baseline, after a 20 session 2-3/w program of physical therapy and at a follow up of 3 months.

The evaluations of the first phase will be implemented with evaluation of mobility and balance using Six Minute Walking Test (6MWT), Mini Balance Evaluation System Test (MiniBESTest) and Timed Up and Go test (TUG).

ELIGIBILITY:
Inclusion Criteria:

* Subject suffering from peripheral neuropathy with a TNSc© score more than 4
* male and female subjects who are 18 years of age or older

Exclusion Criteria:

* orthopedic or neurologic comorbidities that can influence postural control

A control group of healthy subjects with the same demographic features of peripheral neuropathy patients wil be also included.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Peripheral neuropathy patients sent for a neurologic evaluation
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of multi-muscle synergy organization using Synergy Index (SI) | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Multi-muscle Synergy Index (SI) are new measurements of postural stability and a proxy of multi-muscle coordination. Synergy has been defined as a neural organization of a large set of effectors (e.g., muscles) providing stability of salient performance variables (e.g., center of pressure, COP). Within this framework, SI has been introduced, reflecting the relative amount of inter-trial variance that does not affect a performance variable.
Evaluation of change in Anticipatory Synergy Adjustments (ASA) | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  ASAs represent changes in an index of a multi-muscle synergy stabilizing the coordinate of the center of pressure (COP). Such changes may be seen in young, healthy persons about 200-300 ms prior to the action initiation.
Evaluation of balance | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of balance using Mini Balance Evaluation System Test (MiniBESTest). Each item is scored on a 0-4 scale; the scores are summed to obtain a total score of 28. The item are divided in four sessions: anticipatory, reactive postural control, sensory orientation, dynamic gait.
Evaluation of balance | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of balance using Timed Up and Go test (TUG). It is a measure of the time taken by the patient for rising from a chair, walking three meters, turning and walking back to the chair to sit down.
Evaluation of mobility | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of mobility using Six Minute Walking Test (6MWT). The 6MWT assesses distance walked over six minutes as a sub-maximal test of endurance/aerobic capacity.

SECONDARY OUTCOMES:
Severity of chemotherapy induced-peripheral neuropathy | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Total Neuropathy Score-clinical version (TNSc©)
Evaluation of change in electromyography (EMG) parameters | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of sensory conduction velocity of ulnar, radial and sural nerves.
Evaluation of change in electromyography (EMG) parameters | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of motory conduction velocity of ulnar, radial and peroneal nerves.
Impact of PN on patients' quality of life | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of quality of life using the Short Form Health Survey 36 (SF-36). It is a self-report measure of functional health and well-being. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items).
Evaluation of change in level of disability | At baseline, after the 20th session of the rehabilitation program, follow up at 3 months
  Evaluation of level of disability using Functional Independence Measure (FIM). It is an 18-item, seven-level, ordinal scale intended to be sensitive to changes over the course of a comprehensive inpatient medical rehabilitation program.It includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Paola ALberti, MD, PhD, Principal Investigator — Università degli Studi di Milano Bicocca; Cecilia Perin, MD, Principal Investigator — Università degli Studi di Milano Bicocca; Guido Cavaletti, MD, Study Director — Università degli Studi di Milano Bicocca
Locations (2):
- Italy (2):
  - Cecilia Perin, Carate Brianza, Monza E Brianza
  - Paola Alberti, Monza, Monza E Brianza

IPD SHARING:
Plan to Share IPD: Undecided